CLINICAL TRIAL: NCT01531621
Title: A Population-based Prospective Study to Evaluate Clinical Behaviour, Resectability and Survival in 1st Line Metastatic Colorectal Cancer (CRC) Patients in Finland
Brief Title: A Population-based Prospective Study of Metastatic Colorectal Cancer (CRC) Patients in Finland
Acronym: RAXO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pia Osterlund (Other)
Responsible Party: Sponsor-Investigator, Pia Osterlund, Principal Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Other Study IDs: 2011-003158-24
Record Dates: First submitted 2012-02-03; First posted 2012-02-13 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mCRC treatments: All used treatments for metastatic colorectal cancer
  Interventions: Other: Biomarker sampling

INTERVENTIONS:
Other: Biomarker sampling — Blood samples every 8-12 weeks

SUMMARY:
* A population-based prospective study to evaluate clinical behaviour, resectability and survival in 1st line metastatic colorectal cancer (CRC) patients in Finland
* Primary objective: To assess clinical behaviour of metastatic colorectal cancer and overall resectability, postoperative morbidity and outcomes after resection
* Secondary objectives: To assess treatments for mCRC; To assess efficacy of chemotherapy and targeted drugs with overall response rates (ORR), failure free survival (FFS), progression free survival (PFS), and overall survival (OS); To radiologically assess tumour density and morphology, and assess alternative radiologic response evaluation in comparison with RECIST response criteria; To evaluate whole blood, plasma, serum and tumour block biomarkers and DNA polymorphisms that may predict drug effects, resectability and clinical behaviour of the tumour

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed CRC, who are scheduled to start or are getting first line chemotherapy for metastatic disease
2. Age > 18
3. Metastatic disease (including locally advanced disease not amenable with surgery and/or (chemo)radiotherapy)
4. Signed written informed consent according to ICH/GCP and the local regulations (approved by the Independent Ethics Committee [IEC]) will be obtained prior to study
5. No informed consent will be obtained from patients participating in the data collection study obtaining data from hospital charts. No blood sampling, nor contacting of patients will be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic cancer of the colon or rectum
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-02; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Resectability | 5 years
  To assess clinical behaviour of metastatic colorectal cancer and overall resectability, postoperative morbidity and outcomes after resection

SECONDARY OUTCOMES:
Efficacy | 5 years
  Response rates
Safety | 5 years
  Number of adverse events
Radiological assessment | 5 years
  To radiologically assess tumour density and morphology, and assess alternative radiologic response evaluation in comparison with RECIST response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pia Osterlund, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Department of Oncology, Helsinki, Finland

REFERENCES:
- [Derived] Uutela A, Osterlund E, Halonen P, Kallio R, Algars A, Salminen T, Lamminmaki A, Soveri LM, Ristamaki R, Lehtomaki K, Stedt H, Heerva E, Muhonen T, Kononen J, Nordin A, Ovissi A, Kytola S, Keinanen M, Sundstrom J, Nieminen L, Makinen MJ, Kuopio T, Ristimaki A, Isoniemi H, Osterlund P. Resectability, conversion, metastasectomy and outcome according to RAS and BRAF status for metastatic colorectal cancer in the prospective RAXO study. Br J Cancer. 2022 Sep;127(4):686-694. doi: 10.1038/s41416-022-01858-8. Epub 2022 May 24. PMID 35610367
- [Derived] Uutela A, Ovissi A, Hakkarainen A, Ristimaki A, Lundbom N, Kallio R, Soveri LM, Salminen T, Algars A, Halonen P, Ristamaki R, Nordin A, Blanco Sequeiros R, Rinta-Kiikka I, Lantto E, Virtanen J, Paakko E, Liukkonen E, Saunavaara J, Ryymin P, Lammentausta E, Osterlund P, Isoniemi H; RAXO Study Group. Treatment response of colorectal cancer liver metastases to neoadjuvant or conversion therapy: a prospective multicentre follow-up study using MRI, diffusion-weighted imaging and 1H-MR spectroscopy compared with histology (subgroup in the RAXO trial). ESMO Open. 2021 Aug;6(4):100208. doi: 10.1016/j.esmoop.2021.100208. Epub 2021 Jul 26. PMID 34325107